CLINICAL TRIAL: NCT01399775
Title: Evaluation of Implant Stability and Dimensional Changes in Alveolar Ridge Following Immediate Implantation
Brief Title: Evaluation of Ridge Dimensional Changes After Immediate Implantation and Efficacy of This Procedure
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Amir Moeintaghavi, associate professor of periodontics, Mashhad University of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 87703
Record Dates: First submitted 2011-07-21; First posted 2011-07-22 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Atrophy of Edentulous Alveolar Ridge; Alveolar Ridge Augmentation
Keywords: Atrophy of Edentulous Alveolar Ridge; Dental Prosthesis, Implant-Supported; Dental Implants, Single-Tooth
MeSH Terms: interventions — Drug Implants; Embryo Implantation, Delayed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- immediate implantation (Experimental): Immediately after tooth extraction, dental implant is inserted.
  Interventions: Procedure: immediate implantation
- Delayed implantation (Other): Four months after extraction, Dental implant is inserted.
  Interventions: Procedure: Delayed implantation

INTERVENTIONS:
Procedure: immediate implantation — Immediately after tooth extraction, a dental implant is inserted
  Other Names: Implant in fresh socket
  Arms: immediate implantation
Procedure: Delayed implantation — Four months after extraction, a dental implant is inserted and measurements are recorded.
  Arms: Delayed implantation

SUMMARY:
1. Evaluation of dimensional changes in alveolar ridge following immediate implantation compared to delayed implantation
2. evaluation of the effect of gap dimensions between socket walls and dental implant in implant stability

DETAILED DESCRIPTION:
24 hopeless single root teeth will be selected. The horizontal and vertical measurements will be assessed in 12socket after immediate implantation and filling the gape with DFDBA.

Horizontal dimensions (bucco-lingual) of alveolar ridge will be measured at 1,3 and 7 mm using caliper and CBCT , and vertical ridge dimensions at 8 points:(mid-buccal,mid-lingual,mesial,distal,disto-buccal-mesio-buccal,disto-lingual,mesio-lingual ) will be determined using a periodontal probe from the line connecting the two adjacent CEJs ,and dimensional changes will be measured after 3 months following implant insertion with the same device during the second stage surgery.

The vertical and horizontal dimensions between the implant and alveolar crest and between the crest and base of the gap will be measured at 8 points:(mid-buccal,mid-lingual,mesial,distal,disto-buccal-mesio-buccal,disto-lingual,mesio-lingual ).

The primary and secondary stability will be measured using Osstell at baseline and 3-month later.

Twelve sockets will heal without grafting materials, soft and hard tissue measurements including horizontal and vertical ridge dimensions will be determined. All the measurement will be assessed using caliper and CBCT at the time of extraction and 3-month later at the time of implant insertion.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hopeless single root tooth and willing for dental implants
* Having no systemic disease

Exclusion Criteria:

* Fail to osseointegrate

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-05; Primary Completion 2010-12 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
dimensional changes | baseline to 3 months
  Horizontal dimensions (bucco-linguall) of alveolar ridge will be measured at 1,3 and 7 mm using caliper and CBCT , and vertical ridge dimensions at 8 points:(mid-buccal,mid-lingual,mesial,distal,disto-buccal-mesio-buccal,disto-lingual,mesio-lingual ) will be determined using a periodontal probe from the line connecting the two adjacent CEJs ,and dimensional changes will be measured after 3 months following implant insertion with the same device during the second stage surgery.

SECONDARY OUTCOMES:
implant stability | baseline to 3 months
  The primary and secondary stability will be measured using osstell at baseline and 3-month later.

CONTACTS AND LOCATIONS:
Overall Officials: Mehrdad Radvar, DDS., Phd, Study Chair — Mashhad University of Medical Sciences
Locations (1):
- Mashhad University of Medical Sciences, Dental school, Mashhad, Khorasan Razavi, Iran